CLINICAL TRIAL: NCT02123199
Title: Prospective Observational Study of the Impact of Indacaterol (Onbrez®) on the Individual Lives and Health Status of Patients With COPD
Brief Title: Study of the Impact of Indacaterol (Onbrez®) on the Individual Lives and Health Status of Patients With COPD
Acronym: INHALE
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CQAB149BGB01
Record Dates: First submitted 2014-04-22; First posted 2014-04-25 (Estimated); Last update posted 2014-04-25 (Estimated); Status verified 2014-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — indacaterol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Indacaterol/QAB149: Patients treated with Indacaterol for COPD prior to enrollment in study
  Interventions: Drug: Indacaterol (Onbrez®) /QAB149

INTERVENTIONS:
Drug: Indacaterol (Onbrez®) /QAB149

SUMMARY:
A prospective observational multi centre research study in GP practices clustered within up to 10 UK Primary care trusts.

ELIGIBILITY:
Inclusion Criteria:

* Patients with active diagnosis of COPD, confirmed by spirometry documented in medical notes

Exclusion Criteria:

* Patients who are currently receiving other maintenance therapy (except LAMA) for COPD.
* Patients previously prescribed Indacaterol.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be recruited only after indacaterol has been prescribed and is being used for the patients first maintenance therapy for COPD symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2012-04; Primary Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change in COPD assessment Test (CAT Score) at 6-8 weeks after the initiation of indacaterol | 6-8 weeks

SECONDARY OUTCOMES:
Change in COPD Assessment test (CAT) score at 6 months after the initiation of indacaterol | 6 months
Impact of indacaterol on patients' lies at 6 - 8 weeks after the initiation of indacaterol. | 6-8 weeks
Physician Global Evaluation of Treatment effectiveness (GETE) at 6-8 weeks and 6 months. | 6-8 weeks and 6 months
Patient Global Evaluation of Treatment effectiveness (GETE) at 6 months | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, London, London, United Kingdom